CLINICAL TRIAL: NCT01382082
Title: Assessment of Cognitive Function in Breast Cancer and Lymphoma Patients Receiving Chemotherapy at Pre-Treatment, Post-Treatment, at Six Month Follow-Up, and Long-Term Follow-Ups
Brief Title: Assessment of Cognitive Function in Breast Cancer and Lymphoma Patients Receiving Chemotherapy
Acronym: CANTAB
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle Janelsins, PhD, MPH, Professor of Surgery, Radiation Oncology, and Neuroscience, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Other Study IDs: URCC-10055; UG1CA189961 (NIH); U10CA037420 (NIH); NCT01330225 (obsolete NCT alias)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Lymphoma
Keywords: cognitive function; memory; attention; breast cancer; lymphoma
MeSH Terms: conditions — Breast Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- subjects with breast cancer
- subjects with lymphoma
- subjects without cancer

SUMMARY:
Cognitive impairments in cancer patients represent an important clinical problem. Studies to date estimating prevalence of difficulties in memory, executive function, and attention deficits have been limited by small sample sizes and many have lacked healthy control groups. More information is needed on promising biomarkers and allelic variants that may help to determine the etiology of impairment, identify those most vulnerable to impairment, and develop interventions for these difficulties.

This is a longitudinal observational study of cognitive function in breast cancer and lymphoma patients receiving chemotherapy to better understand the prevalence of cognitive difficulties (i.e., problems with memory, executive function, and attention) in these populations.

ELIGIBILITY:
Inclusion Criteria:

Subjects Receiving Chemotherapy:

* Have a diagnosis of invasive breast cancer (stage I-IIIC) or intermediate or high-grade* lymphoma (*defined by the treating physician)
* Be scheduled to begin a course of chemotherapy
* Oral chemotherapy is acceptable
* Previous or concurrent treatment with hormones or biological response modifiers is acceptable. (Subjects receiving biological response modifiers only are not eligible).
* Be chemotherapy naïve
* Life expectancy greater than 10 months
* Be able to speak and read English
* Give written informed consent

Inclusion Criteria, Controls:

* Must be the same gender as the subject receiving chemotherapy
* Must be within 5 years of the age of the subject receiving chemotherapy
* Life expectancy greater than 10 months
* Be able to speak and read English
* Give written informed consent
* Must be willing to participate in the study for the entire period

Inclusion Criteria, Long-Term Followup Study:

* Must be a subject who had breast cancer, or control who was paired with that subject with breast cancer, who provided CANTAB data at any time-point during assessments 1 through 3.

Exclusion Criteria:

Subjects Receiving Chemotherapy:

* Must not be currently hospitalized or have been hospitalized within the last year for a psychiatric illness
* Must not be diagnosed with a neurodegenerative disease
* Must not have primary central nervous system (CNS) disease
* Must not have received chemotherapy in the past
* Must not be scheduled to receive concurrent radiation treatment
* Must not have metastatic disease (subjects with breast cancer)
* Must not be pregnant
* Must not be colorblind

Exclusion Criteria, Controls:

* Must not be currently hospitalized or have been hospitalized within the last year for a psychiatric illness
* Must not be diagnosed with a neurodegenerative disease
* Must not have primary CNS disease
* Must not have been diagnosed with cancer or previously have received chemotherapy
* Must not be pregnant or plan on becoming pregnant during the study period
* Must not be colorblind

Exclusion Criteria, Long-Term Followup Study:

* Must not have dementia or any severe neurodegenerative disease that would prohibit the ability to complete cognitive testing.
* Must not be colorblind

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: During enrollment, the groups will be balanced on age and gender. Controls of the same age and gender as the subject receiving chemotherapy will be enrolled at the same time.
Sampling Method: Non-Probability Sample
Enrollment: 1432 (Estimated)
Dates: Start 2011-07-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short-term memory | Longitudinal Mixed Model assessing change over time from pre to post chemotherapy and at 6 month follow-up assessing change from pre to post chemotherapy and pre to 6 months post-chemotherapy in patients compared to controls
  Change in Short-term visual memory will be assessed by the computerized Delayed Matching to Sample (DMS) task.

SECONDARY OUTCOMES:
Attention impairment | Longitudinal Mixed Model assessing change over time from pre to post chemotherapy and at 6 month follow-up assessing change from pre to post chemotherapy and pre to 6 months post-chemotherapy in patients compared to controls
  Change in attention will be assessed by the computerized Rapid Visual Information Processing (RVP) task.
Verbal recognition memory impairment | Longitudinal Mixed Model assessing change over time from pre to post chemotherapy and at 6 month follow-up assessing change from pre to post chemotherapy and pre to 6 months post-chemotherapy in patients compared to controls
  Change in Memory (verbal) will be assessed by the computerized Verbal Recognition Memory (VRM) Task.
Executive function impairment | Longitudinal Mixed Model assessing change over time from pre to post chemotherapy and at 6 month follow-up assessing change from pre to post chemotherapy and pre to 6 months post-chemotherapy in patients compared to controls
  Change in Executive function will be assessed by the computerized One Touch Stockings of Cambridge (OTS) planning task.
Self-report score | Longitudinal Mixed Model assessing change over time from pre to post chemotherapy and at 6 month follow-up assessing change from pre to post chemotherapy and pre to 6 months post-chemotherapy in patients compared to controls
  FACT-Cog change score
short term memory | 8 and/or 10 years post-chemotherapy
  Delayed match to sample score
attention | 8 and/or 10 years post-chemotherapy
  Rapid Visual Processing speed score
Self-report score | 8 and/or 10 years post-chemotherapy
  FACT-Cog

OTHER OUTCOMES:
correlation of cognitive function with TNF alpha pathway biomarkers | change from pre to post chemotherapy and six month follow up
  serum assaying the change in the TNF pathway

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C. Janelsins, PhD, Study Chair — University of Rochester
Locations (29):
- United States (29):
  - Delaware/Christiana Care NCORP, Newark, Delaware
  - Delaware/Christiana Care NCORP (CHRISTIANA), Newark, Delaware
  - Heartland, Decatur, Illinois
  - Kansas City Clinical Oncology Program, Prairie Village, Kansas
  - Wichita NCORP, Wichita, Kansas
  - Wichita, Wichita, Kansas
  - Gulf South MU-NCORP, New Orleans, Louisiana
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - CRCWM, Grand Rapids, Michigan
  - Metro Minnesota NCORP, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada, Las Vegas, Nevada
  - Hem Onc CNY, East Syracuse, New York
  - Kansas City, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Novant Health Cancer Institute - Kernersville, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Program, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Columbus, Columbus, Ohio
  - Dayton Community Oncology Program, Dayton, Ohio
  - Dayton, Dayton, Ohio
  - Pacific Cancer Research Consortium Ncorp, Portland, Oregon
  - PCRC, Portland, Oregon
  - NCORP of the Carolinas, Greenville, South Carolina
  - Upstate Carolina, Spartanburg, South Carolina
  - Northwest (Virginia Mason), Seattle, Washington
  - Wisconsin NCORP, Marshfield, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kleckner AS, Kleckner IR, Culakova E, Shayne M, Belcher EK, Gudina AT, Williams AM, Onitilo AA, Hopkins JO, Gross H, Mustian KM, Peppone LJ, Janelsins MC. The association between cancer-related fatigue and diabetes from pre-chemotherapy to 6 months post-chemotherapy. Support Care Cancer. 2022 Sep;30(9):7655-7663. doi: 10.1007/s00520-022-07189-x. Epub 2022 Jun 9. PMID 35678881
- [Derived] Gilmore N, Mohile S, Lei L, Culakova E, Mohamed M, Magnuson A, Loh KP, Maggiore R, Belcher E, Conlin A, Weiselberg L, Ontko M, Janelsins M. The longitudinal relationship between immune cell profiles and frailty in patients with breast cancer receiving chemotherapy. Breast Cancer Res. 2021 Feb 5;23(1):19. doi: 10.1186/s13058-021-01388-w. PMID 33546731